CLINICAL TRIAL: NCT00807625
Title: Mucosal and Systemic Responses to Contraceptives in HIV-Infected Women in Zambia
Brief Title: Impact of Different Contraceptives on the Immune System of HIV Infected Women in Zambia
Acronym: MSRC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: F071227004
Record Dates: First submitted 2008-12-11; First posted 2008-12-12 (Estimated); Last update posted 2012-07-13 (Estimated); Status verified 2012-07

CONDITIONS: HIV; Contraception; HIV Infections
Keywords: HIV/AIDS; Contraception; Birth control; CD4+; Viral Load; T-cell activation; B-cell activation; Hormonal; Intrauterine device; Depo Provera; Women; IUCD; treatment naive
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Medroxyprogesterone Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IUCD (Active Comparator): Assigned to use a copper intrauterine device
  Interventions: Device: Copper T Intrauterine contraception device
- DMPA (Active Comparator): Assigned to use Depo Provera
  Interventions: Drug: Depo Provera

INTERVENTIONS:
Drug: Depo Provera — Depo Provera administered by injection at randomization visit and the 12-week study visit.
  Arms: DMPA
Device: Copper T Intrauterine contraception device — IUCD inserted upon randomization to this study arm
  Other Names: ParaGuard TCu 380A
  Arms: IUCD

SUMMARY:
In this study, 66 HIV-infected women who desire contraception will be randomly assigned to use either an IUD or Depo Provera, and will be followed for six months. The study is intended to help investigators understand potential mechanisms by which hormonal contraception may hasten HIV disease progression.

DETAILED DESCRIPTION:
In this randomized controlled trial, 66 HIV-infected women who desire contraception will be assigned to one of two treatment groups: IUD or Depo Provera. The study builds on findings from a previous study which examined the safety and acceptability of hormonal contraception and IUD among HIV-infected women. Secondary analyses from the previous study indicated that women who were assigned to the hormonal arm appeared to have faster disease progression based on death and decline in CD4+ count as compared to women assigned to the IUD arm. With the current study, investigators seek to understand potential mechanisms for the effect of hormonal contraception on hastening HIV disease progression. Enrolled women will be asked to use the assigned contraception method for a period of six months, and various indicators of disease progression will be collected at four follow-up visits after randomization.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed HIV status by local rapid test algorithm
* Willingness to be randomized to a contraceptive method and continue that method for at least 6 months.
* Intention to stay in the study area for at least 6 months

Exclusion Criteria:

* Currently pregnant or pregnant within the prior 6 months
* Currently breastfeeding
* Documented liver disease
* History of coagulation disorder
* Active tuberculosis
* Anemia, defined as Hgb <8gm/dL
* Age < 16 years (the age of consent in Zambia);
* Eligible for antiretroviral therapy based on Zambian National Guidelines (CD4+ < 200, or WHO stage IV, or CD4+< 350 and WHO stage III)
* Currently using an IUD or hormonal method of contraception, or have used a hormonal contraceptive in the past 6 months

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2008-11; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
T-cell activation | 4, 8, 12, and 24 weeks post-randomization

SECONDARY OUTCOMES:
CD4+ cell decline | 4, 8, 12, and 24 weeks post-randomization
Cervical viral load | 4, 8, 12, and 24 weeks post-randomization

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth M Stringer, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- The Centre for Infectious Disease Research in Zambia, Lusaka, Lusaka Province, Zambia